CLINICAL TRIAL: NCT03439839
Title: An Open Label, Single Arm, Multiple Dose Study to Assess Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of LNP023 When Administered in Addition to Standard of Care (SoC) in Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH) With Signs of Active Hemolysis
Brief Title: Study of Safety, Efficacy, Tolerability, Pharmacokinetics and Pharmacodynamics of LNP023 in in Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLNP023X2201; 2017-000888-33 (EudraCT Number)
Record Dates: First submitted 2018-02-14; First posted 2018-02-20 (Actual); Results first posted 2024-01-03 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH) With Signs of Active Hemolysis
Keywords: Complement; alternative pathway; paroxysmal nocturnal hemoglobinuria; hemolysis
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal; Hemolysis | interventions — iptacopan; Standard of Care

STUDY DESIGN:
Intervention Model Description: Open label, non-randomized study
Masking Description: No masking used in the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: LNP023 200mg bid + SoC (Experimental): Orally administered iptacopan 200 mg b.i.d. in Part 1 and Part 2
  Interventions: Drug: iptacopan; Combination Product: Standard of Care
- Cohort 2: LNP023 50mg/200mg bid + SoC (Experimental): Orally administered iptacopan 50 mg b.i.d. for a minimum of 2 weeks in addition to SoC; this could be increased to iptacopan 200 mg b.i.d. at study day 15 or at any time later in the study if LDH was not within limit of normal or reduced by at least 60% as compared to baseline values.
  Interventions: Drug: iptacopan; Combination Product: Standard of Care

INTERVENTIONS:
Drug: iptacopan — iptacopan bid orally administered
  Other Names: LNP023
Combination Product: Standard of Care — Standard of Care (SoC) is defined as an antibody with anti C5 activity. At the time of study start, eculizumab was the only available SoC; eculizumab will be hereafter referred to as SoC.

SUMMARY:
This was a Phase 2, open label, single arm, multiple dose study to assess efficacy, safety, pharmacokinetics and pharmacodynamics of iptacopan when administered in addition to Standard of care (SoC) in patients with paroxysmal nocturnal hemoglobinuria (PNH) with signs of active hemolysis.

DETAILED DESCRIPTION:
LNP023 is a novel oral small molecular weight compound that inhibits factor B (FB) of the alternative pathway (AP). Blockade of the AP with oral LNP023 has the potential to prevent both intra - and extravascular hemolysis.

This two-cohort study consisted of a screening period of up to 68 days, a baseline visit, and Treatment periods Part 1 and Part 2. The planned duration of Treatment Part 1 was 13 weeks; the planned duration of Treatment Part 2 (treatment extension for patients who benefit from LNP023 treatment in Part 1 of the study based on reduced hemolytic parameters) was between approximately 2 to 3 years.

Cohort 1: Orally administered iptacopan 200 mg b.i.d. in Part 1 and Part 2 in addition to SoC.

Cohort 2: Orally administered iptacopan 50 mg b.i.d. for a minimum of 2 weeks in addition to SoC; this could be increased to iptacopan 200 mg b.i.d. at study day 15 or at any time later in the study if LDH was not within limit of normal or reduced by at least 60% as compared to baseline values.

End of Study (EoS) visit happened 2 weeks after last LNP023 administration for patients not joining the roll over extension program (REP).

A safety follow-up call was conducted 30 days after last administration of study treatment (applicable only for patients not joining the REP).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients between the age of 18-80 (inclusive) at Baseline with a diagnosis of PNH based on documented clone size of ≥10% by RBCs and/or granulocytes, measured by glycosylphosphatidylinositol (GPI)-deficiency on flow cytometry (screening or medical history data acceptable).
2. For Cohort 1 only: LDH values ≥1.5 × Upper limit of normal (ULN) range for at least 3 pre-SoC dosing measurements taken in relation to 3 different SoC dosing dates over a maximum of 10 weeks prior to Day 1 (Screening, Baseline, or medical history data acceptable). All other Screening pre-SoC LDH values must be >1 × ULN range (for pre-SoC samples collected at the same day as SoC administration).
3. For Cohort 2 only: LDH values ≥1.25 × ULN range for at least 3 pre-SoC dosing measurements taken in relation to 3 different SoC dosing dates over a maximum of 10 weeks prior to Day 1 (Screening, Baseline, or medical history data acceptable). All other Screening pre-SoC LDH values must be >1 × ULN range (for pre-SoC samples collected at the same day as SoC administration).
4. For Cohort 2 only: Hemoglobin level <10.5 g/dL at Baseline.
5. PNH patients on stable regimen of SoC complement blockade (monoclonal antibody with anti C5 activity) for at least 3 months prior to first treatment with iptacopan.
6. Previous vaccination against N. meningitidis types A, C, Y and W-135 is required at least 4 weeks prior to first dosing with iptacopan. Vaccination against N. meningitidis type B should be conducted if available and acceptable by local regulations, at least 4 weeks prior to first dosing with iptacopan. If iptacopan treatment must start earlier than 4 weeks post vaccination, prophylactic antibiotic treatment must be initiated.
7. Previous vaccination for the prevention of S. pneumoniae and H. influenzae at least 4 weeks prior to first dosing with iptacopan. If iptacopan treatment must start earlier than 4 weeks post vaccination, prophylactic antibiotic treatment must be initiated.

Exclusion Criteria:

1. Known or suspected hereditary complement deficiency at Screening.
2. History of hematopoietic stem cell transplantation as verified both at Screening and at Baseline (unless baseline was skipped).
3. Patients with laboratory evidence of bone marrow failure.
4. A positive Human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C test result at Screening.
5. Presence or suspicion (based on judgment of the Investigator) of active infection within 2 weeks prior to first dose of iptacopan, or history of severe recurrent bacterial infections.
6. History of recurrent meningitis, history of meningococcal infections despite vaccination as verified both at Screening and at Baseline (unless Baseline was skipped).
7. Patients on immunosuppressive agents such as (but not limited to) cyclosporine, mycophenolate mofetil, tacrolimus, cyclophosphamide, methotrexate less than 8 weeks prior to first treatment with iptacopan unless on a stable regimen for at least 3 months prior to first iptacopan dose.
8. Systemic corticosteroids administered at the dose of ≥10 mg per day prednisone equivalent within less than 4 weeks prior to first treatment with iptacopan.
9. Severe concurrent co-morbidities; e.g., patients with severe kidney disease (dialysis), advanced cardiac disease (New York Heart disease Association (NYHA) class IV), severe pulmonary arterial hypertension (World Health Organization (WHO) class IV), unstable thrombotic event not amenable to active treatment as judged by the Investigator both at Screening and at Baseline (unless Baseline was skipped).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Novartis Investigative Site, Paris, France
- Novartis Investigative Site, Essen, Germany
- Novartis Investigative Site, Napoli, Italy

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Result] Risitano AM, Roth A, Soret J, Frieri C, de Fontbrune FS, Marano L, Alashkar F, Benajiba L, Marotta S, Rozenberg I, Milojevic J, End P, Nidamarthy PK, Junge G, Peffault de Latour R. Addition of iptacopan, an oral factor B inhibitor, to eculizumab in patients with paroxysmal nocturnal haemoglobinuria and active haemolysis: an open-label, single-arm, phase 2, proof-of-concept trial. Lancet Haematol. 2021 May;8(5):e344-e354. doi: 10.1016/S2352-3026(21)00028-4. Epub 2021 Mar 23. PMID 33765419
- See also: Patient Lay Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1440

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 3 investigative sites in 3 countries: France (1), Italy (1) and Germany (1).
Pre-assignment Details: All patients needed to complete vaccinations against N. meningitidis, S. pneumoniae and H. influenzae at least 4 weeks prior to starting LNP023 treatment. If LNP023 treatment had to start earlier than 4 weeks post vaccination, prophylactic antibiotic treatment was initiated. Prior to treatment, both cohorts underwent a screening period of up to 68 days followed by a baseline visit.
Groups:
- Cohort 1: LNP023 200mg Bid + SoC: Orally administered iptacopan 200 mg b.i.d. in Part 1 and Part 2 in addition to SoC.
Period: Overall Study
Arm/Group | Cohort 1: LNP023 200mg Bid + SoC | Cohort 2: LNP023 50mg/200mg Bid + SoC
Started | 10 | 6
Completed | 7 | 6
Not Completed | 3 | 0
Not completed — Death | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: LNP023 200mg Bid + SoC | Cohort 2: LNP023 50mg/200mg Bid + SoC | Total
Number analyzed (Participants) | 10 | 6 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 6 | 15
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (15.57) | 51.7 (9.83) | 47.1 (13.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 7 | 3 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Unknown | 0 | 1 | 1
  White | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Lactate Dehydrogenase (LDH) Level at Day 92
Description: Serum LDH was used as an intravascular hemolysis marker to assess the effect of iptacopan on the reduction of chronic hemolysis in paroxysmal nocturnal hemoglobinuria (PNH) patients when administered in addition to SoC (monoclonal antibody with anti C5 activity)
  Baseline is defined as the mean of the last 3 measurements prior to dose administration.
Time Frame: Baseline and Day 92
Population: The Pharmacodynamic (PD) analysis set is defined as patients with available PD data and no protocol deviations with relevant impact on PD data.
  The overall number of participants analyzed represents the participants in the PD analysis set who had valid measurements of LDH at Baseline and Day 92.
Measure: Mean (90% Confidence Interval); unit: Percent change from Baseline
Groups:
- Total: Participants from Cohort 1 and Cohort 2
Arm/Group | Cohort 1: LNP023 200mg Bid + SoC | Cohort 2: LNP023 50mg/200mg Bid + SoC | Total
Number analyzed (Participants) | 9 | 5 | 14
Percent change from Baseline | -53.59 [-61.38 to -45.79] | -25.56 [-46.92 to -4.20] | -43.58 [-53.57 to -33.58]

2. Secondary Outcome: Absolute Change From Baseline in Lactate Dehydrogenase (LDH) Level
Description: as for outcome 1
Time Frame: Baseline, day 8, 15, 29, 57 and 92
Population: The overall number of participants analyzed represents the participants in the PD analysis set.
  The number analyzed per row represents the participants with a valid LDH value at both baseline and that particular visit
Measure: Mean (90% Confidence Interval); unit: U/L
Arm/Group | Cohort 1: LNP023 200mg Bid + SoC | Cohort 2: LNP023 50mg/200mg Bid + SoC | Total
Number analyzed (Participants) | 10 | 6 | 16
U/L
  Day 8 | -272.57 [-349.07 to -196.07] | -145.22 [-196.30 to -94.15] | -224.81 [-279.88 to -169.74]
  Day 15: number analyzed (Participants) | 10 | 5 | 15
  Day 15 | -353.97 [-486.36 to -221.57] | -175.07 [-247.55 to -102.59] | -294.33 [-388.42 to -200.24]
  Day 29 | -368.17 [-510.15 to -226.18] | -191.22 [-258.88 to -123.56] | -301.81 [-395.89 to -207.73]
  Day 57 | -317.07 [-459.11 to -175.03] | -135.89 [-212.28 to -59.50] | -249.13 [-344.24 to -154.01]
  Day 92: number analyzed (Participants) | 9 | 5 | 14
  Day 92 | -330.52 [-488.02 to -173.01] | -109.07 [-196.69 to -21.45] | -251.43 [-361.88 to -140.98]

3. Secondary Outcome: Absolute Change From Baseline in Hemoglobin
Description: Hemoglobin was used as a marker of intra and extravascular hemolysis when administered in addition to SoC (monoclonal antibody with anti C5 activity) to assess the effect of iptacopan.
  Baseline is defined as the mean of all pre-dose measurements.
Time Frame: Baseline; day 1, 2, 8, 15, 22, 29, 36, 43, 57, 71, 85, 92, 113, 127, 141, 155, 169, 197, 225, 253, 281, 309, 337, 393, 449, 505, 561, 617, 673, 729, 785, 841, 897, 953, 1009, 1065, 1121, 1177, 1233
Population: The overall number of participants analyzed represents the participants in the PD analysis set.
  The number analyzed per row represents the participants with a valid hemoglobin value at both baseline and that particular visit.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Cohort 1: LNP023 200mg Bid + SoC | Cohort 2: LNP023 50mg/200mg Bid + SoC
Number analyzed (Participants) | 10 | 6
g/L
  Day 1: number analyzed (Participants) | 10 | 5
  Day 1 | -4.05 (8.750) | -6.67 (7.218)
  Day 2 | -3.65 (7.638) | -8.06 (6.830)
  Day 8 | 12.85 (9.228) | 20.11 (13.475)
  Day 15 | 20.25 (10.122) | 26.44 (10.047)
  Day 22 | 24.15 (11.898) | 35.11 (11.065)
  Day 29 | 28.25 (13.131) | 35.11 (10.141)
  Day 36 | 29.55 (12.166) | 33.94 (10.062)
  Day 43 | 26.15 (12.571) | 31.11 (7.428)
  Day 57 | 27.05 (10.855) | 35.94 (10.804)
  Day 71: number analyzed (Participants) | 8 | 4
  Day 71 | 24.53 (12.259) | 28.54 (8.080)
  Day 85: number analyzed (Participants) | 10 | 3
  Day 85 | 28.65 (15.722) | 30.72 (15.008)
  Day 92: number analyzed (Participants) | 10 | 5
  Day 92 | 31.85 (14.543) | 32.43 (14.584)
  Day 113: number analyzed (Participants) | 9 | 5
  Day 113 | 30.14 (14.831) | 32.43 (11.092)
  Day 127: number analyzed (Participants) | 9 | 4
  Day 127 | 33.92 (16.882) | 38.92 (13.519)
  Day 141: number analyzed (Participants) | 10 | 5
  Day 141 | 28.05 (17.088) | 37.23 (15.802)
  Day 155: number analyzed (Participants) | 8 | 5
  Day 155 | 28.28 (17.370) | 37.83 (12.287)
  Day 169: number analyzed (Participants) | 10 | 5
  Day 169 | 27.05 (17.253) | 39.43 (11.174)
  Day 197: number analyzed (Participants) | 10 | 3
  Day 197 | 28.95 (15.429) | 31.89 (16.385)
  Day 225: number analyzed (Participants) | 10 | 3
  Day 225 | 28.65 (17.258) | 28.67 (7.147)
  Day 253: number analyzed (Participants) | 10 | 4
  Day 253 | 26.95 (18.015) | 28.17 (12.039)
  Day 281: number analyzed (Participants) | 9 | 4
  Day 281 | 29.91 (18.351) | 45.54 (16.168)
  Day 309: number analyzed (Participants) | 9 | 4
  Day 309 | 27.17 (15.152) | 36.29 (9.866)
  Day 337: number analyzed (Participants) | 9 | 4
  Day 337 | 26.28 (16.733) | 32.50 (10.700)
  Day 393: number analyzed (Participants) | 9 | 4
  Day 393 | 28.47 (18.801) | 39.79 (12.930)
  Day 449: number analyzed (Participants) | 8 | 5
  Day 449 | 31.22 (18.573) | 37.93 (10.547)
  Day 505: number analyzed (Participants) | 7 | 6
  Day 505 | 24.89 (13.435) | 44.28 (18.271)
  Day 561: number analyzed (Participants) | 6 | 5
  Day 561 | 29.25 (18.665) | 40.13 (11.653)
  Day 617: number analyzed (Participants) | 7 | 6
  Day 617 | 32.23 (18.335) | 42.78 (17.771)
  Day 673: number analyzed (Participants) | 5 | 5
  Day 673 | 38.42 (13.407) | 38.13 (15.418)
  Day 729: number analyzed (Participants) | 8 | 4
  Day 729 | 31.28 (15.366) | 34.92 (11.357)
  Day 785: number analyzed (Participants) | 4 | 4
  Day 785 | 11.63 (22.691) | 40.04 (26.752)
  Day 841: number analyzed (Participants) | 7 | 4
  Day 841 | 24.27 (18.109) | 38.54 (23.649)
  Day 897: number analyzed (Participants) | 7 | 2
  Day 897 | 31.85 (17.303) | 56.83 (20.035)
  Day 953: number analyzed (Participants) | 6 | 0
  Day 953 | 23.93 (14.964) |
  Day 1009: number analyzed (Participants) | 7 | 0
  Day 1009 | 23.99 (19.396) |
  Day 1065: number analyzed (Participants) | 6 | 0
  Day 1065 | 29.07 (17.334) |
  Day 1121: number analyzed (Participants) | 7 | 0
  Day 1121 | 27.27 (14.536) |
  Day 1177: number analyzed (Participants) | 5 | 0
  Day 1177 | 32.28 (11.180) |
  Day 1233: number analyzed (Participants) | 5 | 0
  Day 1233 | 33.08 (10.196) |

4. Secondary Outcome: Absolute Change From Baseline in Free Hemoglobin
Description: Free hemoglobin was used as a marker of intra and extravascular hemolysis when administered in addition to SoC (monoclonal antibody with anti C5 activity) to assess the effect of iptacopan.
  Baseline is defined as the mean of all pre-dose measurements.
Time Frame: as for outcome 3
Population: The overall number of participants analyzed represents the participants in the PD analysis set.
  The number analyzed per row represents the participants with a valid free hemoglobin value at both baseline and that particular visit.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cohort 1: LNP023 200mg Bid + SoC | Cohort 2: LNP023 50mg/200mg Bid + SoC
Number analyzed (Participants) | 10 | 6
mg/dL
  Day 1 | 15.26 (36.879) | 9.16 (15.310)
  Day 2 | -26.73 (40.706) | -3.94 (6.785)
  Day 8: number analyzed (Participants) | 9 | 6
  Day 8 | -24.03 (43.102) | -2.04 (6.725)
  Day 15 | -23.16 (41.190) | 14.21 (43.762)
  Day 22 | -22.90 (39.726) | -0.66 (6.960)
  Day 29 | -20.03 (42.349) | -1.21 (8.108)
  Day 36 | -12.42 (47.495) | -2.56 (6.914)
  Day 43: number analyzed (Participants) | 9 | 6
  Day 43 | -13.63 (24.961) | -0.54 (6.546)
  Day 57: number analyzed (Participants) | 8 | 6
  Day 57 | 1.71 (14.138) | -1.84 (6.662)
  Day 71: number analyzed (Participants) | 9 | 4
  Day 71 | -17.92 (34.378) | 0.18 (1.466)
  Day 85: number analyzed (Participants) | 10 | 4
  Day 85 | -16.80 (47.407) | 1.90 (2.338)
  Day 92: number analyzed (Participants) | 8 | 5
  Day 92 | -25.12 (42.237) | -3.31 (6.295)
  Day 113: number analyzed (Participants) | 9 | 5
  Day 113 | -24.00 (41.084) | 16.09 (42.454)
  Day 127: number analyzed (Participants) | 9 | 5
  Day 127 | -18.07 (52.791) | 1.42 (2.945)
  Day 141: number analyzed (Participants) | 10 | 5
  Day 141 | -24.03 (40.625) | -1.52 (8.137)
  Day 155: number analyzed (Participants) | 9 | 4
  Day 155 | -20.58 (43.690) | -2.43 (8.741)
  Day 169: number analyzed (Participants) | 9 | 5
  Day 169 | -1.00 (91.222) | 10.24 (19.275)
  Day 197: number analyzed (Participants) | 10 | 4
  Day 197 | 14.93 (105.958) | 3.19 (5.185)
  Day 225: number analyzed (Participants) | 10 | 3
  Day 225 | 10.64 (101.866) | 15.89 (32.159)
  Day 253: number analyzed (Participants) | 10 | 4
  Day 253 | -21.97 (40.320) | 34.84 (61.838)
  Day 281: number analyzed (Participants) | 10 | 5
  Day 281 | -24.19 (39.910) | -1.36 (7.326)
  Day 309: number analyzed (Participants) | 10 | 4
  Day 309 | -21.57 (42.638) | -2.26 (9.656)
  Day 337: number analyzed (Participants) | 9 | 3
  Day 337 | -20.69 (42.592) | 31.39 (55.947)
  Day 393: number analyzed (Participants) | 9 | 3
  Day 393 | -17.29 (42.263) | -2.11 (8.297)
  Day 449: number analyzed (Participants) | 8 | 5
  Day 449 | -28.60 (44.210) | -3.93 (7.781)
  Day 505: number analyzed (Participants) | 7 | 6
  Day 505 | -33.24 (41.787) | -1.69 (6.335)
  Day 561: number analyzed (Participants) | 7 | 4
  Day 561 | -34.25 (43.692) | 1.59 (2.372)
  Day 617: number analyzed (Participants) | 7 | 5
  Day 617 | -34.68 (44.127) | -0.22 (6.960)
  Day 673: number analyzed (Participants) | 5 | 4
  Day 673 | -37.43 (54.005) | 2.39 (15.832)
  Day 729: number analyzed (Participants) | 8 | 4
  Day 729 | -28.88 (38.550) | -3.99 (7.294)
  Day 785: number analyzed (Participants) | 4 | 2
  Day 785 | -2.55 (4.388) | -0.67 (3.206)
  Day 841: number analyzed (Participants) | 7 | 4
  Day 841 | -33.12 (43.462) | 1.60 (4.485)
  Day 897: number analyzed (Participants) | 4 | 2
  Day 897 | -12.98 (22.233) | 4.77 (5.468)
  Day 953: number analyzed (Participants) | 7 | 0
  Day 953 | -34.41 (46.196) |
  Day 1009: number analyzed (Participants) | 7 | 0
  Day 1009 | 8.39 (135.082) |
  Day 1065: number analyzed (Participants) | 7 | 0
  Day 1065 | -34.10 (44.867) |
  Day 1121: number analyzed (Participants) | 7 | 0
  Day 1121 | -33.45 (43.628) |
  Day 1177: number analyzed (Participants) | 3 | 0
  Day 1177 | -16.30 (23.441) |
  Day 1233: number analyzed (Participants) | 3 | 0
  Day 1233 | -12.27 (20.734) |

5. Secondary Outcome: Absolute Change From Baseline in Reticulocytes Count
Description: Reticulocytes count was used as a marker of intra and extravascular hemolysis when administered in addition to SoC (monoclonal antibody with anti C5 activity) to assess the effect of iptacopan.
  Baseline is defined as the mean of all pre-dose measurements.
Time Frame: as for outcome 3
Population: The overall number of participants analyzed represents the participants in the PD analysis set.
  The number analyzed per row represents the participants with a valid reticulocyte count value both at baseline and that particular visit
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Cohort 1: LNP023 200mg Bid + SoC | Cohort 2: LNP023 50mg/200mg Bid + SoC
Number analyzed (Participants) | 10 | 6
10^9 cells/L
  Day 1: number analyzed (Participants) | 10 | 5
  Day 1 | 4.44 (33.269) | 1.62 (22.790)
  Day 2 | 8.61 (52.306) | 4.39 (31.658)
  Day 8 | -96.94 (69.179) | -104.55 (88.085)
  Day 15 | -130.15 (80.335) | -130.40 (107.295)
  Day 22 | -139.26 (78.206) | -147.70 (99.438)
  Day 29 | -132.28 (76.822) | -169.68 (129.743)
  Day 36 | -130.73 (72.017) | -167.51 (137.214)
  Day 43 | -129.02 (64.301) | -160.05 (132.859)
  Day 57 | -117.69 (65.394) | -149.53 (116.803)
  Day 71: number analyzed (Participants) | 8 | 4
  Day 71 | -106.83 (62.973) | -146.87 (129.217)
  Day 85: number analyzed (Participants) | 10 | 5
  Day 85 | -113.96 (65.278) | -167.16 (156.013)
  Day 92: number analyzed (Participants) | 10 | 5
  Day 92 | -110.54 (62.638) | -150.02 (105.893)
  Day 113: number analyzed (Participants) | 9 | 6
  Day 113 | -96.78 (66.366) | -147.06 (129.118)
  Day 127: number analyzed (Participants) | 9 | 4
  Day 127 | -107.84 (57.904) | -149.92 (115.401)
  Day 141: number analyzed (Participants) | 10 | 5
  Day 141 | -115.17 (70.942) | -108.39 (54.412)
  Day 155: number analyzed (Participants) | 8 | 5
  Day 155 | -99.90 (62.273) | -98.67 (65.700)
  Day 169: number analyzed (Participants) | 10 | 5
  Day 169 | -109.39 (63.159) | -84.57 (64.082)
  Day 197: number analyzed (Participants) | 10 | 3
  Day 197 | -98.87 (85.280) | -152.09 (137.856)
  Day 225: number analyzed (Participants) | 10 | 3
  Day 225 | -104.11 (72.206) | -143.68 (149.716)
  Day 253: number analyzed (Participants) | 10 | 4
  Day 253 | -104.30 (64.401) | -139.05 (127.212)
  Day 281: number analyzed (Participants) | 9 | 4
  Day 281 | -111.11 (60.896) | -121.06 (66.564)
  Day 309: number analyzed (Participants) | 9 | 4
  Day 309 | -116.88 (51.145) | -114.06 (77.982)
  Day 337: number analyzed (Participants) | 9 | 4
  Day 337 | -113.31 (61.144) | -170.89 (142.577)
  Day 393: number analyzed (Participants) | 9 | 4
  Day 393 | -58.54 (152.003) | -183.20 (122.298)
  Day 449: number analyzed (Participants) | 8 | 5
  Day 449 | -89.44 (77.782) | -152.66 (124.244)
  Day 505: number analyzed (Participants) | 7 | 6
  Day 505 | -100.68 (64.132) | -135.80 (117.488)
  Day 561: number analyzed (Participants) | 6 | 5
  Day 561 | -101.63 (67.525) | -163.34 (121.860)
  Day 617: number analyzed (Participants) | 7 | 6
  Day 617 | -101.73 (54.916) | -132.40 (122.940)
  Day 673: number analyzed (Participants) | 5 | 5
  Day 673 | -137.05 (63.373) | -150.14 (130.898)
  Day 729: number analyzed (Participants) | 8 | 4
  Day 729 | -101.16 (63.442) | -179.15 (131.007)
  Day 785: number analyzed (Participants) | 4 | 4
  Day 785 | -56.22 (26.739) | -134.60 (141.947)
  Day 841: number analyzed (Participants) | 7 | 4
  Day 841 | -103.96 (60.469) | -145.80 (140.363)
  Day 897: number analyzed (Participants) | 7 | 2
  Day 897 | -111.41 (58.641) | -81.27 (36.298)
  Day 953: number analyzed (Participants) | 5 | 0
  Day 953 | -91.00 (52.203) |
  Day 1009: number analyzed (Participants) | 7 | 0
  Day 1009 | -110.33 (61.354) |
  Day 1065: number analyzed (Participants) | 6 | 0
  Day 1065 | -127.35 (61.501) |
  Day 1121: number analyzed (Participants) | 7 | 0
  Day 1121 | -115.96 (55.981) |
  Day 1177: number analyzed (Participants) | 5 | 0
  Day 1177 | -140.14 (73.898) |
  Day 1233: number analyzed (Participants) | 5 | 0
  Day 1233 | -123.40 (70.558) |

6. Secondary Outcome: Absolute Change From Baseline in C3 Fragment Deposition on PNH RBC
Description: C3 fragment deposition on PNH Red blood cell (RBC) was used as a marker of intra and extravascular hemolysis when administered in addition to SoC (monoclonal antibody with anti C5 activity) to assess the effect of iptacopan.
  Baseline is defined as Day 1 pre-dose measurement.
Time Frame: Day 1 pre dose, day 8, 22, 29, 57, 92, 113, 141, 169, 253, 337, 505, 673, 785, 953, 1121, 1233
Population: The overall number of participants analyzed represents the participants in the PD analysis set who had at least one valid measurement of C3 fragment deposition.
  The number analyzed per row represents the participants with a valid C3 fragment deposition value both at baseline and that particular visit
Measure: Mean (Standard Deviation); unit: percentage of PNH RBC
Arm/Group | Cohort 1: LNP023 200mg Bid + SoC | Cohort 2: LNP023 50mg/200mg Bid + SoC
Number analyzed (Participants) | 10 | 5
percentage of PNH RBC
  Day 8 | -5.59 (6.541) | -1.24 (4.510)
  Day 22: number analyzed (Participants) | 8 | 4
  Day 22 | -8.02 (8.198) | -2.35 (5.620)
  Day 29: number analyzed (Participants) | 8 | 5
  Day 29 | -11.64 (7.990) | -4.36 (2.662)
  Day 57: number analyzed (Participants) | 8 | 3
  Day 57 | -8.90 (5.778) | -5.35 (2.357)
  Day 92: number analyzed (Participants) | 7 | 3
  Day 92 | -8.70 (6.310) | -6.21 (0.866)
  Day 113: number analyzed (Participants) | 7 | 2
  Day 113 | -13.65 (9.927) | -5.10 (2.478)
  Day 141: number analyzed (Participants) | 6 | 2
  Day 141 | -13.18 (11.489) | -6.19 (4.818)
  Day 169: number analyzed (Participants) | 7 | 2
  Day 169 | -11.06 (5.874) | -4.66 (3.175)
  Day 253: number analyzed (Participants) | 9 | 4
  Day 253 | -10.08 (6.259) | -4.36 (1.538)
  Day 337: number analyzed (Participants) | 7 | 2
  Day 337 | -11.21 (6.118) | -4.08 (3.340)
  Day 505: number analyzed (Participants) | 3 | 4
  Day 505 | -16.04 (2.732) | -6.76 (2.650)
  Day 673: number analyzed (Participants) | 4 | 0
  Day 673 | -15.19 (2.805) |
  Day 785: number analyzed (Participants) | 1 | 0
  Day 785 | -1.00 |
  Day 953: number analyzed (Participants) | 2 | 0
  Day 953 | -15.28 (3.528) |
  Day 1121: number analyzed (Participants) | 1 | 0
  Day 1121 | -0.94 |
  Day 1233: number analyzed (Participants) | 1 | 0
  Day 1233 | -12.74 |

7. Secondary Outcome: Mean PNH Clone Size
Description: Mean PNH clone size on Red Blood Cells (RBC) was used as a marker of intra and extravascular hemolysis when administered in addition to SoC (monoclonal antibody with anti C5 activity) to assess the effect of iptacopan.
  Baseline is defined as the mean of all pre-dose measurements.
Time Frame: Day 1 pre dose, day 8, 22, 29, 57, 92, 113, 141, 169, 253, 337, 505, 673, 785, 953, 1121, 1233
Population: The overall number of participants analyzed represents the participants in the PD analysis set.
  The number analyzed per row represents the participants with a valid clone size value for that particular visit.
Measure: Mean (Standard Deviation); unit: percentage of PNH RBC
Arm/Group | Cohort 1: LNP023 200mg Bid + SoC | Cohort 2: LNP023 50mg/200mg Bid + SoC
Number analyzed (Participants) | 10 | 6
percentage of PNH RBC
  Day 1 pre dose: number analyzed (Participants) | 10 | 5
  Day 1 pre dose | 54.75 (32.536) | 46.10 (31.436)
  Day 8: number analyzed (Participants) | 9 | 6
  Day 8 | 66.32 (29.570) | 64.45 (27.711)
  Day 22: number analyzed (Participants) | 8 | 5
  Day 22 | 75.23 (23.458) | 79.37 (20.270)
  Day 29: number analyzed (Participants) | 8 | 6
  Day 29 | 75.34 (20.837) | 78.87 (17.642)
  Day 57: number analyzed (Participants) | 9 | 5
  Day 57 | 85.87 (15.660) | 86.45 (12.576)
  Day 92: number analyzed (Participants) | 8 | 5
  Day 92 | 89.20 (16.861) | 85.38 (12.939)
  Day 113: number analyzed (Participants) | 8 | 3
  Day 113 | 89.28 (18.936) | 86.02 (9.626)
  Day 141: number analyzed (Participants) | 8 | 3
  Day 141 | 93.91 (6.105) | 80.25 (6.638)
  Day 169: number analyzed (Participants) | 8 | 3
  Day 169 | 87.60 (19.644) | 83.69 (11.187)
  Day 253: number analyzed (Participants) | 9 | 4
  Day 253 | 90.30 (18.176) | 82.28 (12.649)
  Day 337: number analyzed (Participants) | 8 | 3
  Day 337 | 88.69 (20.381) | 91.68 (11.905)
  Day 505: number analyzed (Participants) | 3 | 5
  Day 505 | 98.33 (1.738) | 88.45 (10.419)
  Day 673: number analyzed (Participants) | 4 | 2
  Day 673 | 97.45 (2.370) | 92.48 (6.626)
  Day 785: number analyzed (Participants) | 2 | 0
  Day 785 | 83.61 (9.327) |
  Day 953: number analyzed (Participants) | 2 | 0
  Day 953 | 96.08 (3.825) |
  Day 1121: number analyzed (Participants) | 2 | 0
  Day 1121 | 93.74 (7.410) |
  Day 1233: number analyzed (Participants) | 3 | 0
  Day 1233 | 69.83 (43.045) |

8. Secondary Outcome: Mean Haptoglobin Levels
Description: Haptoglobin level was used as a marker of intra and extravascular hemolysis when administered in addition to SoC (monoclonal antibody with anti C5 activity) to assess the effect of iptacopan.
  Baseline is defined as the mean of all pre-dose measurements.
Time Frame: Day 2, 8, 15, 22, 29, 36, 43, 57, 71, 85, 92, 113, 127, 141, 155, 169, 197, 225, 253, 281, 309, 337, 393, 449, 505, 561, 617, 673, 729, 785, 841, 897, 953, 1009, 1065, 1121, 1177, 1233
Population: The overall number of participants analyzed represents the participants in the PD analysis set.
  The number analyzed per row represents the participants with a valid haptoglobin value for that particular visit.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Cohort 1: LNP023 200mg Bid + SoC | Cohort 2: LNP023 50mg/200mg Bid + SoC
Number analyzed (Participants) | 9 | 4
g/L
  Day 2: number analyzed (Participants) | 2 | 2
  Day 2 | 0.55 (0.071) | 0.30 (0.141)
  Day 8: number analyzed (Participants) | 7 | 3
  Day 8 | 0.70 (0.548) | 0.77 (0.306)
  Day 15: number analyzed (Participants) | 9 | 2
  Day 15 | 0.93 (0.960) | 0.60 (0.141)
  Day 22: number analyzed (Participants) | 8 | 4
  Day 22 | 1.18 (1.387) | 0.70 (0.483)
  Day 29: number analyzed (Participants) | 7 | 3
  Day 29 | 0.94 (0.896) | 0.83 (0.586)
  Day 36: number analyzed (Participants) | 5 | 3
  Day 36 | 1.08 (0.779) | 0.97 (0.503)
  Day 43: number analyzed (Participants) | 5 | 3
  Day 43 | 1.26 (1.401) | 0.70 (0.520)
  Day 57: number analyzed (Participants) | 3 | 1
  Day 57 | 0.63 (0.416) | 1.20
  Day 71: number analyzed (Participants) | 4 | 1
  Day 71 | 0.75 (0.473) | 0.80
  Day 85: number analyzed (Participants) | 3 | 0
  Day 85 | 0.87 (0.611) |
  Day 92: number analyzed (Participants) | 2 | 1
  Day 92 | 0.95 (0.495) | 0.80
  Day 113: number analyzed (Participants) | 3 | 1
  Day 113 | 0.63 (0.493) | 0.50
  Day 127: number analyzed (Participants) | 3 | 0
  Day 127 | 0.47 (0.208) |
  Day 141: number analyzed (Participants) | 3 | 1
  Day 141 | 0.57 (0.306) | 0.70
  Day 155: number analyzed (Participants) | 1 | 1
  Day 155 | 0.50 | 0.80
  Day 169: number analyzed (Participants) | 3 | 1
  Day 169 | 0.63 (0.577) | 0.50
  Day 197: number analyzed (Participants) | 3 | 0
  Day 197 | 0.80 (0.700) |
  Day 225: number analyzed (Participants) | 4 | 0
  Day 225 | 0.65 (0.705) |
  Day 253: number analyzed (Participants) | 4 | 0
  Day 253 | 0.63 (0.519) |
  Day 281: number analyzed (Participants) | 2 | 1
  Day 281 | 0.50 (0.283) | 0.30
  Day 309: number analyzed (Participants) | 2 | 1
  Day 309 | 0.75 (0.071) | 0.50
  Day 337: number analyzed (Participants) | 1 | 0
  Day 337 | 0.40 |
  Day 393: number analyzed (Participants) | 2 | 0
  Day 393 | 0.60 (0.283) |
  Day 449: number analyzed (Participants) | 1 | 1
  Day 449 | 0.20 | 0.60
  Day 505: number analyzed (Participants) | 2 | 1
  Day 505 | 0.60 (0.141) | 0.60
  Day 561: number analyzed (Participants) | 1 | 1
  Day 561 | 0.60 | 0.70
  Day 617: number analyzed (Participants) | 2 | 2
  Day 617 | 0.30 (0.141) | 1.90 (1.838)
  Day 673: number analyzed (Participants) | 1 | 1
  Day 673 | 0.30 | 0.70
  Day 729: number analyzed (Participants) | 2 | 1
  Day 729 | 0.35 (0.071) | 0.50
  Day 785: number analyzed (Participants) | 1 | 2
  Day 785 | 1.00 | 1.25 (0.919)
  Day 841: number analyzed (Participants) | 3 | 2
  Day 841 | 0.47 (0.153) | 0.85 (0.212)
  Day 897: number analyzed (Participants) | 3 | 0
  Day 897 | 0.33 (0.058) |
  Day 953: number analyzed (Participants) | 2 | 0
  Day 953 | 0.50 (0.141) |
  Day 1009: number analyzed (Participants) | 2 | 0
  Day 1009 | 0.45 (0.071) |
  Day 1065: number analyzed (Participants) | 2 | 0
  Day 1065 | 2.05 (1.768) |
  Day 1121: number analyzed (Participants) | 4 | 0
  Day 1121 | 1.00 (0.935) |
  Day 1177: number analyzed (Participants) | 2 | 0
  Day 1177 | 0.40 (0.000) |
  Day 1233: number analyzed (Participants) | 2 | 0
  Day 1233 | 0.95 (0.636) |

9. Secondary Outcome: Absolute Change From Baseline in Total Bilirubin
Description: Bilirubin was used as a marker of intra and extravascular hemolysis when administered in addition to SoC (monoclonal antibody with anti C5 activity) to assess the effect of iptacopan.
  Baseline is defined as the mean of all pre-dose measurements.
Time Frame: as for outcome 3
Population: The overall number of participants analyzed represents the participants in the PD analysis set.
  The number analyzed per row represents the participants with a valid bilirubin value both at baseline and that particular visit.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Cohort 1: LNP023 200mg Bid + SoC | Cohort 2: LNP023 50mg/200mg Bid + SoC
Number analyzed (Participants) | 10 | 6
umol/L
  Day 1 | 2.94 (13.038) | 1.36 (4.978)
  Day 2 | -21.06 (15.647) | -25.47 (21.598)
  Day 8 | -23.66 (16.081) | -25.97 (24.380)
  Day 15 | -23.86 (16.538) | -26.97 (24.043)
  Day 22 | -25.36 (15.403) | -25.14 (23.541)
  Day 29 | -24.66 (15.026) | -26.14 (22.345)
  Day 36 | -23.96 (15.945) | -25.31 (27.658)
  Day 43 | -24.66 (14.552) | -25.14 (23.727)
  Day 57 | -24.16 (13.946) | -22.81 (21.233)
  Day 71: number analyzed (Participants) | 10 | 4
  Day 71 | -23.16 (15.154) | -27.92 (24.924)
  Day 85: number analyzed (Participants) | 10 | 4
  Day 85 | -23.66 (14.595) | -28.42 (26.075)
  Day 92: number analyzed (Participants) | 10 | 5
  Day 92 | -21.66 (13.985) | -27.87 (25.234)
  Day 113: number analyzed (Participants) | 9 | 5
  Day 113 | -21.06 (15.026) | -26.87 (23.200)
  Day 127: number analyzed (Participants) | 9 | 4
  Day 127 | -22.18 (13.357) | -27.79 (26.965)
  Day 141: number analyzed (Participants) | 10 | 5
  Day 141 | -22.46 (14.404) | -18.23 (9.473)
  Day 155: number analyzed (Participants) | 9 | 5
  Day 155 | -19.73 (12.376) | -16.23 (9.565)
  Day 169: number analyzed (Participants) | 10 | 5
  Day 169 | -21.66 (13.383) | -14.83 (10.281)
  Day 197: number analyzed (Participants) | 9 | 4
  Day 197 | -24.21 (13.678) | -23.71 (28.849)
  Day 225: number analyzed (Participants) | 10 | 3
  Day 225 | -23.06 (12.410) | -30.06 (36.183)
  Day 253: number analyzed (Participants) | 10 | 4
  Day 253 | -21.36 (12.192) | -24.21 (30.342)
  Day 281: number analyzed (Participants) | 10 | 4
  Day 281 | -23.46 (12.150) | -16.54 (8.694)
  Day 309: number analyzed (Participants) | 10 | 4
  Day 309 | -22.86 (12.078) | -11.21 (10.635)
  Day 337: number analyzed (Participants) | 10 | 4
  Day 337 | -22.76 (13.248) | -28.71 (29.338)
  Day 393: number analyzed (Participants) | 9 | 4
  Day 393 | -19.73 (15.644) | -28.00 (27.769)
  Day 449: number analyzed (Participants) | 8 | 5
  Day 449 | -24.64 (13.021) | -23.50 (25.603)
  Day 505: number analyzed (Participants) | 7 | 6
  Day 505 | -27.30 (12.450) | -25.81 (24.978)
  Day 561: number analyzed (Participants) | 7 | 5
  Day 561 | -21.98 (14.718) | -21.10 (30.888)
  Day 617: number analyzed (Participants) | 6 | 6
  Day 617 | -28.85 (11.516) | -23.47 (21.451)
  Day 673: number analyzed (Participants) | 5 | 5
  Day 673 | -27.58 (13.453) | -24.50 (25.562)
  Day 729: number analyzed (Participants) | 8 | 4
  Day 729 | -23.64 (12.971) | -32.13 (28.799)
  Day 785: number analyzed (Participants) | 4 | 4
  Day 785 | -11.54 (5.370) | -26.67 (33.656)
  Day 841: number analyzed (Participants) | 7 | 4
  Day 841 | -20.49 (12.006) | -29.42 (32.316)
  Day 897: number analyzed (Participants) | 7 | 2
  Day 897 | -24.49 (13.627) | -16.00 (7.542)
  Day 953: number analyzed (Participants) | 7 | 0
  Day 953 | -23.92 (14.707) |
  Day 1009: number analyzed (Participants) | 7 | 0
  Day 1009 | -23.92 (14.204) |
  Day 1065: number analyzed (Participants) | 6 | 0
  Day 1065 | -25.65 (13.844) |
  Day 1121: number analyzed (Participants) | 7 | 0
  Day 1121 | -23.35 (14.363) |
  Day 1177: number analyzed (Participants) | 5 | 0
  Day 1177 | -29.78 (11.559) |
  Day 1233: number analyzed (Participants) | 5 | 0
  Day 1233 | -28.78 (12.328) |

10. Secondary Outcome: Number of Participants With on Study Transfusions From Packed RBC Units
Description: Number of participants with on study transfusions from packed RBC units was collected.
Time Frame: Up to 46 months
Population: The overall number of participants analyzed represents the participants in the safety analysis set.
  Safety analysis set included all patients that received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: LNP023 200mg Bid + SoC | Cohort 2: LNP023 50mg/200mg Bid + SoC
Number analyzed (Participants) | 10 | 6
Participants | 2 | 2

11. Secondary Outcome: Pharmacokinetics Profile: Maximum Plasma Concentration (Cmax)
Description: Cmax is the maximum (peak) observed plasma drug concentration after single dose administration (mass x volume-1).
  PK assessment parameters were determined using the actual recorded sampling times and non-compartmental methods.
  In Cohort 2, patients were supposed to be orally administered iptacopan 50 mg b.i.d. in addition to SoC; this was increased to iptacopan 200 mg b.i.d. at study day 15 or at any time later in the study if LDH was not within limit of normal or reduced by at least 60% as compared to baseline values. One patient in Cohort 2 was orally administered iptacopan 25 mg at day 1 due to a dosing error.
Time Frame: Day 1, 29, 169, 337
Population: The overall number of participants analyzed represents the participants in the PK analysis set.
  The Pharmacokinetic (PK) analysis set is defined as patients with at least one available valid PK concentration measurement, who received any study drug and with no protocol deviations that impact on PK data.
  The number analyzed per row represents the participants with a valid Cmax value for that particular visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cohort 2: LNP023 25mg Bid + SoC: Orally administered iptacopan 25 mg b.i.d. at the respective visit due to dosing error
- Cohort 2: LNP023 50mg Bid + SoC: Orally administered iptacopan 50 mg b.i.d. at the respective visit
- Cohort 2: LNP023 200mg Bid + SoC: Orally administered iptacopan 200 mg b.i.d. at the respective visit
Arm/Group | Cohort 1: LNP023 200mg Bid + SoC | Cohort 2: LNP023 25mg Bid + SoC | Cohort 2: LNP023 50mg Bid + SoC | Cohort 2: LNP023 200mg Bid + SoC
Number analyzed (Participants) | 10 | 1 | 6 | 3
ng/mL
  Day 1: number analyzed (Participants) | 10 | 1 | 5 | 0
  Day 1 | 3400 (1060) | 1610 | 1570 (366) |
  Day 29: number analyzed (Participants) | 10 | 0 | 6 | 0
  Day 29 | 3500 (1340) |  | 1770 (469) |
  Day 169: number analyzed (Participants) | 9 | 0 | 1 | 3
  Day 169 | 3530 (853) |  | 1180 | 3130 (824)
  Day 337: number analyzed (Participants) | 9 | 0 | 1 | 3
  Day 337 | 4030 (1140) |  | 2470 | 4370 (1790)

12. Secondary Outcome: Pharmacokinetics Profile: Area Under the Curve (AUC) Tau
Description: The AUCtau is the area under the plasma concentration-time curve calculated to the end of a dosing interval (tau) at steady-state.
  PK assessment parameters were determined using the actual recorded sampling times and non-compartmental methods.
  In Cohort 2, patients were supposed to be orally administered iptacopan 50 mg b.i.d. in addition to SoC; this was increased to iptacopan 200 mg b.i.d. at study day 15 or at any time later in the study if LDH was not within limit of normal or reduced by at least 60% as compared to baseline values. One patient in Cohort 2 was orally administered iptacopan 25 mg at day 1 due to a dosing error.
Time Frame: day 1, 29, 169, 337
Population: The overall number of participants analyzed represents the participants in the PK analysis set.
  The number analyzed per row represents the participants with a valid AUCtau value for that particular visit.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort 1: LNP023 200mg Bid + SoC | Cohort 2: LNP023 25mg Bid + SoC | Cohort 2: LNP023 50mg Bid + SoC | Cohort 2: LNP023 200mg Bid + SoC
Number analyzed (Participants) | 10 | 1 | 6 | 3
h*ng/mL
  Day 1: number analyzed (Participants) | 10 | 1 | 5 | 0
  Day 1 | 18200 (6700) | 9470 | 8620 (1310) |
  Day 29: number analyzed (Participants) | 10 | 0 | 6 | 0
  Day 29 | 24400 (8720) |  | 14800 (4100) |
  Day 169: number analyzed (Participants) | 9 | 0 | 1 | 3
  Day 169 | 25600 (7570) |  | 10700 | 23900 (5920)
  Day 337: number analyzed (Participants) | 9 | 0 | 1 | 3
  Day 337 | 26900 (7640) |  | 16900 | 37800 (15500)

13. Secondary Outcome: Pharmacokinetics Profile: Time to Reach Maximum Plasma Concentration (Tmax)
Description: Tmax is the time to reach maximum (peak) plasma drug concentration after single dose administration (time).
  PK assessment parameters were determined using the actual recorded sampling times and non-compartmental methods.
  In Cohort 2, patients were supposed to be orally administered iptacopan 50 mg b.i.d. in addition to SoC; this was increased to iptacopan 200 mg b.i.d. at study day 15 or at any time later in the study if LDH was not within limit of normal or reduced by at least 60% as compared to baseline values. One patient in Cohort 2 was orally administered iptacopan 25 mg at day 1 due to a dosing error.
Time Frame: Day 1, 29, 169, 337
Population: The overall number of participants analyzed represents the participants in the PK analysis set.
  The number analyzed per row represents the participants with a valid Tmax value for that particular visit.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: LNP023 200mg Bid + SoC | Cohort 2: LNP023 25mg Bid + SoC | Cohort 2: LNP023 50mg Bid + SoC | Cohort 2: LNP023 200mg Bid + SoC
Number analyzed (Participants) | 10 | 1 | 6 | 3
hours
  Day 1: number analyzed (Participants) | 10 | 1 | 5 | 0
  Day 1 | 1.50 [1.00 to 6.00] | 2.00 [2.00 to 2.00] | 2.00 [2.00 to 2.00] |
  Day 29: number analyzed (Participants) | 10 | 0 | 6 | 0
  Day 29 | 2.00 [1.00 to 2.00] |  | 2.04 [2.00 to 4.00] |
  Day 169: number analyzed (Participants) | 9 | 0 | 1 | 3
  Day 169 | 2.00 [1.00 to 4.00] |  | 4.00 [4.00 to 4.00] | 2.00 [1.83 to 2.00]
  Day 337: number analyzed (Participants) | 9 | 0 | 1 | 3
  Day 337 | 2.00 [1.00 to 2.00] |  | 2.03 [2.03 to 2.03] | 2.00 [1.05 to 5.00]

14. Secondary Outcome: Red Blood Cell Count: Mean Erythrocytes Levels
Description: Erythrocytes levels were used as a marker of intra and extravascular hemolysis when administered in addition to SoC (monoclonal antibody with anti C5 activity) to assess the effect of iptacopan.
Time Frame: Screening, Baseline, Day 2,8,15,22,29,36,43,57,71,85,92,113,127,141,155,169,197,225,253,281,309,337,393,449,505,561,617,673,729,729,785,841,897,953,1009,1065,1121,1177,1233
Population: The safety analysis set is defined as patients that received any study drug. The number analyzed per row represents the participants with a valid erythrocytes value for that particular visit
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Cohort 1: LNP023 200mg Bid + SoC | Cohort 2: LNP023 50mg/200mg Bid + SoC
Number analyzed (Participants) | 10 | 6
10^12 cells/L
  Screening: number analyzed (Participants) | 9 | 5
  Screening | 3.12 (0.887) | 2.42 (0.427)
  Baseline: number analyzed (Participants) | 9 | 5
  Baseline | 2.73 (0.466) | 2.40 (0.442)
  Day 1: number analyzed (Participants) | 10 | 5
  Day 1 | 2.67 (0.615) | 2.16 (0.498)
  Day 2 | 2.70 (0.485) | 2.17 (0.520)
  Day 8 | 3.17 (0.585) | 3.00 (0.812)
  Day 15 | 3.43 (0.723) | 3.23 (0.794)
  Day 22 | 3.58 (0.835) | 3.57 (0.900)
  Day 29 | 3.72 (0.857) | 3.62 (0.870)
  Day 36 | 3.75 (0.753) | 3.62 (0.804)
  Day 43 | 3.67 (0.807) | 3.55 (0.758)
  Day 57 | 3.69 (0.852) | 3.72 (0.574)
  Day 71: number analyzed (Participants) | 8 | 4
  Day 71 | 3.50 (0.787) | 3.48 (0.591)
  Day 85: number analyzed (Participants) | 10 | 3
  Day 85 | 3.65 (0.841) | 3.60 (0.520)
  Day 92: number analyzed (Participants) | 10 | 5
  Day 92 | 3.76 (0.828) | 3.56 (0.483)
  Day 113: number analyzed (Participants) | 9 | 5
  Day 113 | 3.58 (0.807) | 3.58 (0.444)
  Day 127: number analyzed (Participants) | 9 | 4
  Day 127 | 3.69 (0.822) | 3.75 (0.265)
  Day 141: number analyzed (Participants) | 10 | 5
  Day 141 | 3.64 (0.799) | 3.44 (0.493)
  Day 155: number analyzed (Participants) | 8 | 5
  Day 155 | 3.53 (0.815) | 3.52 (0.432)
  Day 169: number analyzed (Participants) | 10 | 5
  Day 169 | 3.62 (0.826) | 3.54 (0.378)
  Day 197: number analyzed (Participants) | 10 | 3
  Day 197 | 3.68 (0.774) | 3.77 (0.577)
  Day 225: number analyzed (Participants) | 10 | 3
  Day 225 | 3.70 (0.894) | 3.43 (0.513)
  Day 253: number analyzed (Participants) | 10 | 4
  Day 253 | 3.62 (0.930) | 3.45 (0.412)
  Day 281: number analyzed (Participants) | 9 | 4
  Day 281 | 3.81 (0.875) | 3.73 (0.403)
  Day 309: number analyzed (Participants) | 9 | 4
  Day 309 | 3.50 (0.728) | 3.58 (0.427)
  Day 337: number analyzed (Participants) | 9 | 4
  Day 337 | 3.50 (0.714) | 3.75 (0.580)
  Day 393: number analyzed (Participants) | 9 | 4
  Day 393 | 3.63 (0.876) | 4.00 (0.356)
  Day 449: number analyzed (Participants) | 8 | 5
  Day 449 | 3.80 (0.920) | 3.94 (0.378)
  Day 505: number analyzed (Participants) | 7 | 6
  Day 505 | 3.63 (1.053) | 3.92 (0.360)
  Day 561: number analyzed (Participants) | 6 | 5
  Day 561 | 3.47 (0.937) | 3.92 (0.370)
  Day 617: number analyzed (Participants) | 7 | 6
  Day 617 | 3.80 (1.149) | 3.85 (0.389)
  Day 673: number analyzed (Participants) | 5 | 5
  Day 673 | 3.74 (0.716) | 3.86 (0.270)
  Day 729: number analyzed (Participants) | 8 | 4
  Day 729 | 3.74 (1.021) | 3.93 (0.150)
  Day 785: number analyzed (Participants) | 4 | 4
  Day 785 | 2.83 (0.618) | 3.78 (0.263)
  Day 841: number analyzed (Participants) | 7 | 4
  Day 841 | 3.64 (1.081) | 3.80 (0.294)
  Day 897: number analyzed (Participants) | 7 | 2
  Day 897 | 3.89 (1.123) | 3.95 (0.071)
  Day 953: number analyzed (Participants) | 6 | 0
  Day 953 | 3.62 (1.196) |
  Day 1009: number analyzed (Participants) | 7 | 0
  Day 1009 | 3.61 (1.316) |
  Day 1065: number analyzed (Participants) | 6 | 0
  Day 1065 | 3.87 (1.073) |
  Day 1121: number analyzed (Participants) | 7 | 0
  Day 1121 | 3.69 (1.006) |
  Day 1177: number analyzed (Participants) | 5 | 0
  Day 1177 | 4.06 (0.829) |
  Day 1233: number analyzed (Participants) | 5 | 0
  Day 1233 | 4.14 (0.844) |

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 14 days post treatment, up to a maximum duration of 187 weeks. Serious adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of 189 weeks.
Groups:
- Cohort 2: LNP023 50mg Bid + SoC: Orally administered iptacopan 50 mg b.i.d. in Part 1 and iptacopan 50 mg b.i.d. or 200 mg b.i.d. in Part 2 in addition to SoC.
  This arm summarizes all events that started when treated with iptacopan 50 mg b.i.d. in Cophort 2
- Cohort 2: LNP023 200mg Bid + SoC: Orally administered iptacopan 50 mg b.i.d. in Part 1 and iptacopan 50 mg b.i.d. or 200 mg b.i.d. in Part 2 in addition to SoC.
  This arm summarizes all events that started when treated with iptacopan 200 mg b.i.d. in Cohort 2. Total number at risk only includes patients who received LNP023 200mg bid.
- Total: Total
Arm/Group | Cohort 1: LNP023 200mg Bid + SoC | Cohort 2: LNP023 50mg Bid + SoC | Cohort 2: LNP023 200mg Bid + SoC | Total
All-Cause Mortality (participants affected / at risk) | 3/10 | 0/6 | 0/5 | 3/16
Serious Adverse Events (participants affected / at risk) | 4/10 | 0/6 | 2/5 | 6/16
Other Adverse Events (participants affected / at risk) | 10/10 | 4/6 | 5/5 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: LNP023 200mg Bid + SoC (N=10) | Cohort 2: LNP023 50mg Bid + SoC (N=6) | Cohort 2: LNP023 200mg Bid + SoC (N=5) | Total (N=16)
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 1
Urinary bladder polyp (Renal and urinary disorders) | 0 | 0 | 1 | 1
Penetrating aortic ulcer (Vascular disorders) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: LNP023 200mg Bid + SoC (N=10) | Cohort 2: LNP023 50mg Bid + SoC (N=6) | Cohort 2: LNP023 200mg Bid + SoC (N=5) | Total (N=16)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 3
Palpitations (Cardiac disorders) | 0 | 1 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Tongue ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Asthenia (General disorders) | 2 | 2 | 0 | 4
Chest pain (General disorders) | 1 | 0 | 0 | 1
Medical device site irritation (General disorders) | 1 | 0 | 0 | 1
Medical device site pain (General disorders) | 1 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 3 | 1 | 1 | 5
Hepatic cytolysis (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Ocular icterus (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 1 | 0 | 2
Ear infection (Infections and infestations) | 1 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 1 | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 2
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 1
Periodontitis (Infections and infestations) | 1 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 2 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Vaginal infection (Infections and infestations) | 1 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Foot fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 1
SARS-CoV-2 test negative (Investigations) | 0 | 0 | 1 | 1
Weight decreased (Investigations) | 1 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyperferritinaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Angiofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Ageusia (Nervous system disorders) | 0 | 1 | 0 | 1
Anosmia (Nervous system disorders) | 0 | 1 | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 2 | 2 | 1 | 5
Migraine (Nervous system disorders) | 1 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 1 | 0 | 3
Nightmare (Psychiatric disorders) | 1 | 0 | 0 | 1
Poor quality sleep (Psychiatric disorders) | 1 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 2 | 0 | 1 | 3
Haematuria (Renal and urinary disorders) | 0 | 0 | 2 | 2
Nocturia (Renal and urinary disorders) | 1 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 1 | 2
Urinary bladder polyp (Renal and urinary disorders) | 0 | 0 | 1 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Genital discomfort (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Haematospermia (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 3
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Andropause (Social circumstances) | 1 | 0 | 0 | 1
Flushing (Vascular disorders) | 1 | 0 | 0 | 1
Haematoma (Vascular disorders) | 1 | 1 | 0 | 2
Hot flush (Vascular disorders) | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-07-26): https://cdn.clinicaltrials.gov/large-docs/39/NCT03439839/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/39/NCT03439839/SAP_001.pdf